CLINICAL TRIAL: NCT03556371
Title: Evaluation of N-Acetylcysteine Efficacy to Reduce the Craving and to Prolong THE Abstinence Time of Coca Paste
Brief Title: Evaluation of N-Acetylcysteine Efficacy to Reduce the Craving and to Prolong Abstinence Time of Coca Paste
Acronym: NAC-PBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Concepcion, Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Carmen Betancur, MD, Assistant Professor, University of Concepcion, Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA16I0192
Record Dates: First submitted 2018-04-05; First posted 2018-06-14 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine; Coca Paste; N-Acetylcysteine; Craving; Abstinence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled, phase II-b clinical trial, with a parallel group design with CBP dependent patients in different outpatient care units in the province of Concepción, Chile. Patients who meet the cocaine (CBP) consumption disorder criteria, who have used CBP within the last month and who have started use one year at least prior to admission to the study, will be selected from among the consulting population. Patients who agree to participate in the study must sign an informed consent form before being clinically evaluated. During the evaluations, semi-structured interviews and standardized questionnaires will be used to investigate both consumption habits and symptoms of withdrawal and intensity of CBP craving, among others. All patients in the study will be attended twice weekly to treatment centers for four weeks, reporting craving, possible use of for CBP (as well as urine tests), adverse reactions to the indicated medication, among others.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients admitted will be randomly assigned to one of the two treatment groups, according to the table previously generated by the pharmaceutical chemist (PhCh) of the research team, according to a block randomization system, every 10 patients. This will be done with an Excel spreadsheet of Random Assignment by Blocks delivered by the statistical engineer of the research team to the PhCh to generate a table with patients belonging to both groups and number the bottles with the different treatments to administer according to this. Later, the PhCh will deliver them already numbered to the clinical team, being this clinical team blind to the treatment that each patient will receive (they will only handle the bottles with the number of each patient, without knowing which group each of them will belong to). In addition, both the NAC and the placebo bottles will have the same pharmaceutical presentation, so, the patients will also be blind to the pharmacotherapy they will receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine Treatment (Experimental): Oral administration of two capsules, containing 600 milligrams (mg) of N-acetylcysteine each one, twice day (10.00 and 20.00 hours; Total = 2400 mg/day) for four weeks.
  Interventions: Drug: N-Acetylcysteine
- Placebo oral capsules (Placebo Comparator): Oral administration of two capsules, containing 600 milligrams (mg) of Placebo each one, twice day (10.00 and 20.00 hours; Total = 2400 mg/day) for four weeks.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: N-Acetylcysteine — In each patient recruited, assignation to placebo or N-Acetylcysteine group treatment wil be performed, after he/she has signed the informed consent. In the first visit, the evaluation by the psychiatrist and with the nurse team (structured evaluation, which includes the CCQ-N-10, CSSA, general health evaluation, urine drug test and basal blood screening), will be carried out. The nurse team will supervise the drug intake and they will observe 2 hours late the ADRs and general health status of patient, who will be responsible for the intake of the following medication doses. Each patient will be asked to attend twice week to his/her treatment center, during four weeks and each patient visit the clinical team will record the primary and secondary outcome.
  Other Names: Nacudec; CVE 1340878
  Arms: N-acetylcysteine Treatment
Drug: Placebo oral capsule — In each patient recruited, assignation to placebo or N-Acetylcysteine group treatment wil be performed, after he/she has signed the informed consent. In the first visit, the evaluation by the psychiatrist and with the nurse team (structured evaluation, which includes the CCQ-N-10, CSSA, general health evaluation, urine drug test and basal blood screening), will be carried out. The nurse team will supervise the drug intake and they will observe 2 hours late the ADRs and general health status of patient, who will be responsible for the intake of the following medication doses. Each patient will be asked to attend twice week to his/her treatment center, during four weeks and each patient visit the clinical team will record the primary and secondary outcome.
  Arms: Placebo oral capsules

SUMMARY:
* Introduction: The Cocaine Base Paste (or Coca Paste or CBP), a highly toxic and addictive smokable drug (a by-product of the cocaine extraction chain), has become in the last years a real social scourge for Chile. Today, there is not a pharmacological treatment approved in Chile neither around the world for the management of the withdrawal syndrome nor the dependence caused by the use of this substance. The N-Acetylcysteine (NAC), a derivative of the amino acid cysteine, with mucolytic and antioxidant properties, used in Chile since several years for bronchopulmonary treatments, as well as a hepatic and renal protector, among others, has shown, in animal and human research, that has benefits to reduce the craving for cocaine and in the management of the withdrawal syndrome of this and other psychoactive substances.
* Objectives: To evaluate whether the use of NAC in patients with problematic CBP consumption reduce the craving for this substance and prolong its abstinence time.
* Methods: will be carried out a randomized, double-blind, controlled, phase II-b clinical trial, with a parallel group design with CBP dependent patients in different outpatient care units in the province of Concepción, Chile. Patients who meet the cocaine (CBP) consumption disorder criteria, who have used of CBP within the last month and who have started to use it one year at least prior to admission to the study, will be selected from among the consulting population. Patients who agree to participate in the study must sign an informed consent form before being clinically evaluated. During the evaluations, semi-structured interviews and standardized questionnaires were used to investigate both consumption habits and symptoms of withdrawal and intensity of CBP craving, among others. All patients in the study will be attended twice weekly to treatment centers for four weeks, reporting their craving for CBP, the use of this substance (as well as urine tests), adverse reactions to the indicated medication, among others.
* Expected results: It is expected that, thanks to the use of NAC, patients with CBP use disorder entered to this study significantly reduce their craving to consume this substance, they can prolong the abstinence time of it and they can reduce their falls in CBP consumption.

DETAILED DESCRIPTION:
* Quality assurance plan: With the monitoring of our research through the supervision of the Contract Research Organization named South Cone Alliance.

  * Data checks: With the monitoring of our research through the supervision of the Contract Research Organization named South Cone Alliance.
  * Source data verification: All information of the patients recruited in our study was obtained by the research team directly from each patient, without using to external sources.
  * Data dictionary: None
  * Standard Operating Procedures: Each patient must attend twice a week (every 3 days approximately) to assessment in her/him mental health center with the research team. The interventions are detailed below:
* Number 1 Visit:

  1. Reception by the psychiatrist:

     * Explanation of the nature of the study and signing of informed consent.
     * Clinical evaluation with Semi-Structured Interview and application of MINI.
     * Selection of patients who meet criteria, assignment of the respective entry code to the study and entry to the study with it.
     * Delivery of medicine bottle with the first 28 capsules according to previous randomization (treatment for the 1st week)
  2. Nursing Reception (initial structured evaluation):

     * Application of urine drug test (for detection of cocaine, marijuana, benzodiazepines, opiates, amphetamines.) If positive for opioids, the patient is excluded from this study.
     * Anthropometric evaluation (measure, weigh, BMI)
     * Hemodynamic evaluation (blood pressure (BP), body temperature (BT), heart rate (HR) and breathing rate (BR)) to each patient.
     * Performance of baseline blood test: blood count, glycemia, liver tests and creatininemia.
     * Drug administration.
     * Observation for 2 hours of the patient, in which progress is made in:
     * Application of CCQ-N-10, CSSA and Clinical Global Impression (CGI) scales .
     * Record of adverse reactions / side effects of the medication and
     * Final hemodynamic evaluation (BP, BT, HR, BR).
     * Delivery of card of citations for next assessments (or controls).

     Number 2 Visit:

     Nursing follow-up (follow-up file):
     * Record of Abstinence Days (last use of CBP)
     * Urine drug test application (for cocaine detection).
     * Anthropometric evaluation (measure, weigh, BMI)
     * Hemodynamic evaluation ( BP, BT, HR and BR).
     * Asking about withdrawal symptoms (CSSA application)
     * Asking about craving (VAS-craving and CCQ-N-10 application)
     * Asking about adherence to a treatment: application of Morisky-Green Test
     * UKU Scale Application
     * CGI application.
     * Agreement about time for next assesments (or controls).

     Number 3 Visit: Idem to the number 2 visit more delivery of second medicine bottle with 28 capsules for the second week of treatment by the doctor of the research team.

     Number 4 Visit: Idem to the visit number 2

     Number 5 Visit: Idem to the visit number 2 more delivery of third medicine bottle with 28 capsules for the third week of treatment by the doctor of the research team.

     Number 6 Visit: Idem to the visit number 2

     Number 7 Visit: Idem to the visit number 2 more delivery of fourth medicine bottle with 28 capsules for the fourth week of treatment by the doctor of the research team.

     Number 8 visit: Idem to the visit number 2.

     Number 9 visit: Idem to the visit number 2 more the closing of the study.
     * Sample size assessment: The minimum size necessary for a definitive trial in this case would be 106 subjects calculated according to a power of β = 0.8 to detect at least one effect size of the treatment of d = 0.55 , which corresponds to effect size calculated with data from previous studies with this drug in cocaine-dependent patients (LaRowe y cols. Safety and tolerability of N-acetylcysteine in cocaine-dependent individuals. American Journal on Addictions . 2006: 15(1), 105-110). Considering that the analysis of results would be done through a test more powerful than t for independent samples and a level of significance α = 0.05 will be accepted in a two-tailed design.
     * Plan for missing data:

     First: the missing data pattern will be analyzed Second: The mechanism of missing data will be studied to see if it is possible to predict the loss pattern and evaluate the possible bias for missing data.

     Third: If it is found that the missing data mechanism generates bias, multiple imputation will be used for the analyzes.

     • Statistical analysis plan:

     The main outcomes of this test will be described as follows:
     * the proportion of patients who agreed to enter the trial,
     * the differences between those who entered and those who refused,
     * the characteristics of the sample,
     * adherence to treatment, and
     * the number and characteristics of dropouts during follow-up.
* The characteristics of the participants in each arm of the trial will be compared, but will not be subjected to statistical tests. The variables to be compared will be sex, age, comorbidity, PBC consumption time, severity of CBP use disorder and baseline CBP craving to verify homogeneity between groups.

  * Primary outcomes will be compared at four-week follow-up, as follows:
  * After verifying the distribution of the mean duration of CBP abstinence days in both groups, a model will be analyzed by adjusting according to the severity of the CBP use disorder in the baseline (this is the most relevant variable reported in the literature that could influence to the abstinence) and by adjusting according to previous abstinence days, it means, days without coca paste use before to enter this research.
  * Differences in primary outcome by group (with severity adjustment and previous abstinence days) will be reported along with their 95% confidence intervals.
  * The results will be analyzed using the statistical program SPSS and R. According to the variables of result to be evaluated, the analyzes will be:
  * For tolerability assessment: Proportion comparison test (normal approximation, sample sizes allow) for Adverse Drug Reactions (ADR) for each of the 8 post-basal measurement instances.
  * For safety assessment: proportion of patients with mild, moderate and severe ADR per group analyzed with the Brunner-Munzel test, extension of the Mann-Whitney U for ordinal data with many repetitions.
  * To assess coca paste (CBP) abstinence time: Abstinence days will be compared using a Kaplan-Mier estimator. In the case of finding a signifcant increase in CBP abstinence days in the NAC treatment group, a correlation study (Pearson, if there is normality, Spearman otherwise) will be made between the quantitative variables measured to the individuals and days of abstinence.
  * To evaluate the rate of falls in CBP consumption: Fall rates in CBP consumption will be compared using a generalized linear mixed model, with Poisson response and times between exponential relapses. In case of over-dispersion, a model with Negative Binomial response will be considered.
  * For Craving evaluation: it will be analyzed by means of test comparisons of means (Student T, under normality verified with Kolmogorov Smirnov, or U Mann Whitney, otherwise) for independent samples, considering the initial measurements (before there is much desertion ).
  * A comparison of means between experimental and control groups will be performed using repeated measures ANOVA (if normality is verified with Kolmogorov Smirnov and Fisher homoscedasticity) or non-parametric ANOVA analysis for repeated measures (otherwise).
  * It is also important to mention that incomplete data due to abandonment of the study, whether or not there is a return, should be considered for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* To be a patient asking for treatment in any clinical center participating of our research
* To be 18 years old or older.
* To meet the criteria for cocaine (coca paste / CBP) use disorder according to the DSM-V (Therefore they must have at least one year using this substance)
* To have the CBP as the main drug of consumption.
* To have consumed CBP during the month prior to the start our treatment.
* To have a history of any previous CBP withdrawal symptoms or at the time of admission to the study.
* To accept to participate in this study and to sign informed consent previous to enter to it.

Exclusion Criteria:

* To be pregnant or breastfeeding.
* To have dependence of any substance other than CBP, alcohol, nicotine or marijuana.
* To have a severe alcohol withdrawal syndrome during the study.
* To be a delirium at the time of the study.
* To have a psychiatric disorder that decreases their ability to consent or participate adequately in our study (mental retardation, psychotic disorder, generalized disorder of development or another similar disorder).
* To have an active peptic ulcer.
* To have a active bronchial asthma or severe respiratory disease.
* To have epilepsy or a history of seizures.
* To have a serious medical illness known or in treatment (ex.: cancer, liver or kidney failure).
* To be using drugs such as penicillin, tetracycline, carbamazepine, nitroglycerin, antitussives or inhibitors of bronchial secretion, at the time of the study.
* To have a history of allergy to the NAC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Maximun Number of Cocaine Base Paste (CBP) Abstinence Days During Four weeks | Four weeks
  This outcome will be measured by recording the days without consumption of CBP during the entire duration of the study. This data will be obtained from the report of each patient as well as through the results of urine drug test at each visit of the patient to the treatment center. Finally, we will considered the maximun number of days of CBP abstinence in the 4 weeks of followed of each patient like outcome measure and we will compare the average between both treatment group.

SECONDARY OUTCOMES:
Change From Baseline Craving for Cocaine Base Paste (CBP) at Four Weeks | Four weeks
  This outcome will be measured watching the change from the baseline in the values of Visual Analog Scale for Craving (VAS-Craving) at the 4 weeks.
Relapses Rates According to Arm of Treatment | Four weeks
  We will measure the number of relapses in the CBP consumption of patients in both treatment groups, which will be calculated by counting the number of patients who fall into the consumption of CBP during the time of treatment and the proportion of these in each group.
Change From Baseline Score CCQ-N-10 at Four Weeks | Four weeks
  This outcome will be measured watching the change from the baseline in the values of the Cocaine Craving Questionnaire Now-10 (CCQ-N-10) at the 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen G Betancur, MD/PhD(c), Principal Investigator — Universidad de Concepcion; Benjamín Vicente, MD/PhD, Study Chair — Universidad de Concepcion; Carolina P Gómez, PhD, Study Chair — Universidad de Concepcion; María P Casanova, PhD, Study Chair — Universidad de Concepcion
Locations (5):
- Chile (5):
  - Centro Terapéutico Anün, Coronel, Concepción
  - COSAM Lota, Lota, Concepción
  - COSAM San Pedro de la Paz, San Pedro de la Paz, Concepción
  - Therapeutic Community La Casa Chica, Talcahuano, Concepción
  - Psychiatry Service of Hospital Guillermo Grant Benavente, Concepción

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Informed Consent Form (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03556371/ICF_000.pdf
  • Study Protocol (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03556371/Prot_001.pdf
  • Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03556371/SAP_002.pdf